CLINICAL TRIAL: NCT05882292
Title: A Phase II Study of ABN401 in Advanced Solid Tumors With c-MET Gene Aberration
Brief Title: c-MET Inhibitor in Advanced Solid Tumors With c-MET Gene Aberration
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Minkyu Jung, Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-0093
Record Dates: First submitted 2023-05-11; First posted 2023-05-31 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Neoplasms
Keywords: ABN401; c-MET gene aberration; solid tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: ABN401
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABN401 (Experimental): ABN401 800 mg will be administered orally once daily immediately after a meal [should be within 1 hour post-meal (fed state)] at approximately the same time each day in a 21-day cycle.
  Interventions: Drug: ABN401

INTERVENTIONS:
Drug: ABN401 — ABN401 800 mg will be administered orally once daily immediately after a meal [should be within 1 hour post-meal (fed state)] at approximately the same time each day in a 21-day cycle.
  Other Names: c-MET inhibitor

SUMMARY:
c-MET is a member of the receptor tyrosine kinase (RTK) family. Essential components of signal transduction pathways regulating processes including cell proliferation, differentiation, migration, metabolism, and cell cycle control, RTKs are established targets as treatment strategies for various cancers. c-MET is expressed mainly in epithelial tissues and is subject to dysregulation manifesting as mutations, amplifications, and overexpression. c-MET is implicated in both primary oncogenesis, metastasis and also as a mechanism of drug resistance. c-MET has a high affinity for its naturally occurring ligand, Hepatocyte Growth Factor (HGF, also known as Scatter Factor). Binding of HGF to c-MET induces several complex signaling pathways, resulting in cell proliferation, survival, motility, induction of cells polarity, scattering, angiogenesis, and invasion. c-MET alterations are identified in various cancers.

Several drugs targeting c-MET inhibition have been developed, and capmatinib was approved by FDA in patients with non-small cell lung cancer harboring MET exon 14 skipping mutation. ABN401 competitively attaches to the ATP binding sites in the kinase domain of c-MET with high specificity to inhibit phosphorylation of downstream signaling pathways. Following several animal studies of advanced solid cancers, the first-in-human trial of ABN401 showed anti-tumor activity without DLT, and the phase 2 trial is ongoing.

Recently, the basket trials have been emphasized for tissue agnostic approach targeting certain genetic alterations, and the NCI-MATCH (National Cancer Institute-MATCH) trials in 3,000 patients with advanced solid cancers are ongoing.

Similarly, the KOSMOS-II study is ongoing in Korea. This study is the basket trial that Next-generation sequencing (NGS)-based genetic alterations, which is confirmed in Molecular Tumor Board (MTB), provide the individual treatment approach.

DETAILED DESCRIPTION:
Α. Dose and cycle

- ABN401 800 mg will be administered orally once daily immediately after a meal [should be within 1 hour post-meal (fed state)] at approximately the same time each day in a 21-day cycle.

Β. Treatment duration

* ABN401 will be administered until disease progression, unacceptable toxicity, death, and consent withdrawal.
* Step I: enrolled 8 patients will receive ABN401
* Step II: if more than 3 out of 8 patients showed disease control (complete response, partial response, and stable disease), step II will be forwarded and additional 10 patients will be enrolled.
* If more than 7 out of 18 patients showed disease control, ABN401 will be considered an effective drug in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent for KOSMOS-II master observation study
2. Male or female ≥19 years of age
3. Histologically confirmed advanced solid cancers who harboring c-MET alterations (patients who performed NGS tests and c-MET alterations confirmed in molecular tumor board [MTB]) - exon 14 skipping mutation except for non-small cell lung cancer (NSCLC)

   * c-MET amplification GCN (gene copy no.) ≥6 by NGS
   * Fluorescence/Silver In situ hybridization (FISH/SISH) result of the MET/CEP7 ratio ≥2
   * Other MET alterations that are regarded to be actionable by the KOSMOS MTB
4. Disease progression during or after standard therapy and without further treatment options, or no standard therapy, or ineligible for standard therapy
5. At least one measurable or evaluable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
6. Eastern Cooperative Oncology Group Performance Status 0-2
7. Capable to eat food
8. Adequate organ functions

   * Absolute neutrophil count (ANC) ≥1500/mm3 (ie, 1.5×109/L by International - Unit [IU]); excluding measurements obtained within 7 days after administration of granulocyte colony stimulating factor (G-CSF)
   * Platelet count ≥75000/mm3 (IU: ≥75×109/L); excluding measurements obtained within 7 days after transfusion of platelets.
   * Hemoglobin value of ≥8.0 g/dL
   * AST/ALT ≤3×upper limit of normal (ULN); if liver function abnormalities are due to underlying liver metastasis, AST / ALT ≤5×ULN
   * Total serum bilirubin of ≤1.5×ULN
   * Creatinine clearance (CrCl) of ≥50 mL/min (MDRD)
9. Have a life expectancy of at least 90 days
10. If not menopausal or surgically sterile, willing to practice at least one of the following highly effective methods of birth control for at least a (partner's) menstrual cycle before and for 3 months after study drug administration:

    * Barrier type devices (examples are condom, diaphragm, and contraceptive sponge) used only in combination with a spermicide
    * Sexual intercourse with vasectomized male/sterilized female partner
    * Hormonal female contraceptive (oral, parenteral, intravaginal, implantable, or transdermal) for at least 3 consecutive months prior to investigational product administration (when not clinically contraindicated as in breast, ovarian and endometrial cancers)
    * Use of an intrauterine contraceptive device

      * Note: Abstinence, the rhythm method, and/or contraception by the partner are not acceptable methods of birth control
11. Willing to provide available tissue specimens and consent to blood collection for evaluation of biomarkers

    * Archival tissue specimens: formalin-fixed, paraffin-embedded tissues
    * Optional fresh tissue collection prior to ABN401 administration

Exclusion Criteria:

1. Previous treatment with c-MET inhibitor
2. NSCLC with c-MET exon 14 skipping mutation
3. Previous hypersensitivity reaction to any component of study drugs
4. Presence or history of arrhythmia
5. Past history of

   ① Major surgery within 4 weeks before study (must have complete recovery from surgical complications)

   ② Radiotherapy within 4 weeks before study or limited radiotherapy within 2 weeks

   ③ Chemotherapy or biologic agents within 3 weeks before study (targeted therapy within 2 weeks and mitomycin within 5 weeks)
6. History of the following medical conditions

   * Active central nervous system (CNS) metastasis (clinically unstable after stopping steroid for more than 2 months)
   * Leptomeningeal metastasis
   * Acute systemic infection
   * Acute myocardial infarction, stable/unstable angina, symptomatic heart failure ((New York Heart Association [NYHA] class III or IV within the previous 6 months; if >6 months cardiac function must be within normal limits and the patient must be free of cardiac-related symptoms)
   * Clinically critical chronic vomiting or diarrhea
   * Uncontrolled hypertension (systolic blood pressure >150mmHg diastolic blood pressure>100mmHg)
   * Proteinuria (urine dipstick or 24-hour urine collection > 1.0g): must have 24-hour urine collection if baseline urine dipstick ≥2+
   * Active HBV/ HCV except for

     * HBsAg (+) with undetectable HBV DNA
     * If HBsAg (+) and HBV DNA (+), chronic state of infection and clinically stable after anti-viral therapy for more than 3 months
     * If IgG anti-HBc (+) and past history of HBV infection, undetectable HBV DNA
     * HCV Ab (+) with undetectable HCV RNA
   * Severe psychiatric disorders
   * Concurrent anticoagulants at therapeutic dose
   * Past history of gastrointestinal perforation or fistula within 3 months before study, grade 3 or 4 of gastrointestinal bleeding/varix
7. Toxicity with prior therapy (> grade 1) (except for alopecia, pigmentation, poor oral intake), and neuropathy (> grade 1)
8. Pregnant or breastfeeding
9. Patients with a corrected QT interval (using Fridericia's correction formula) (QTcF) of > 470 msec

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) at 16 weeks | Disease control rate (DCR) at 16 weeks
  Disease control rate (DCR) at 16 weeks

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year
  Overall survival (OS)
Progression-free survival (PFS) | at 16 weeks
  Progression-free survival (PFS)
Objective response rate (ORR) | at 16 weeks
  Objective response rate (ORR)
Duration of response (DoR) | at 16 weeks
  Duration of response (DoR)

CONTACTS AND LOCATIONS:
Overall Officials: minkyu Jung, Principal Investigator — Yonsei Cencer center
Locations (1):
- minkyu Jung, Seoul, Seoul, South Korea